CLINICAL TRIAL: NCT00346190
Title: A Six Month Double-Blind, Placebo-Controlled Trial Followed by Six Month Open-Label Study of the Early Administration of Alendronate on Prevention of Bone Loss After Hip Fracture.
Brief Title: The Study of the Early Administration of Alendronate on Prevention of Bone Loss After Hip Fracture.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CA-16
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2006-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

INTERVENTIONS:
Drug: Alendronate

SUMMARY:
To determine whether administration of Alendronate early is more effective than late in the prevention of osteoporosis following a hip fracture

ELIGIBILITY:
Inclusion Criteria:

Male and Female aged > 55 Low trauma hip fracture up to 90 days Be willing to submit to periodic bone mineral density radiographic studies of the spine & 24 hr urine collection Written informed consent

-

Exclusion Criteria:

* Disorders known to affect bone metabolism Not taking bisphosphonates within last 6 months Drugs known to interfere with calcium metabolism within the lats 6 months prior to hip fracture serum calcium> 2.65 mmol/L Treatment with any investigational drug within the last 30 days

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-01; Study Completion 2007-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kremer, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health center, Montreal, Quebec, Canada